CLINICAL TRIAL: NCT00838266
Title: A Double Blind Randomized, Placebo-controlled, Cross-over Trial to Evaluate the Efficiency of a Mouthrinse, Containing Red Grape Seed Extract and nicométhanol Fluorhydrate, in the Control of Dental Plaque Deposit in a 4-days Plaque Regrowth Model
Brief Title: Study of Growing Biofilm by an Antiplaque Mouthrinse
Acronym: Bain de bouche
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Jean-Pierre LEROY / Clinical Research and Innovation Director, University Hospital, Bordeaux
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CHUBX 2008/05
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Last update posted 2009-09-23 (Estimated); Status verified 2009-09

CONDITIONS: Dental Plaque
Keywords: mouthrinse; grape seed extract; fluor; plaque index
MeSH Terms: conditions — Dental Plaque | interventions — Grape Seed Extract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Antiplaque mouthrinse containing active component (Grape Seed Extract + nicométhanol fluorhydrate)
  Interventions: Drug: mouthrinse (Grape Seed Extract + nicomethanol fluorhydrate)
- 2 (Placebo Comparator): Antiplaque mouthrinse containing non-active component
  Interventions: Other: mouthrinse containing non-active component

INTERVENTIONS:
Drug: mouthrinse (Grape Seed Extract + nicomethanol fluorhydrate) — Antiplaque mouthrinse containing active component three times a day, during 1 minute, for 4 days
  Arms: 1
Other: mouthrinse containing non-active component — Antiplaque mouthrinse containing non-active component three times a day, during 1 minute, for 4 days
  Arms: 2

SUMMARY:
The objective of this study is to evaluate the efficiency of a new mouthrinse on dental plaque deposits.

The study is carried out on 50 volunteers that are asked to use the mouthrinse without any other oral hygiene measure, during 4 days. It is a double bind, cross-over, randomized design: the same subjects test the active product and the placebo.

DETAILED DESCRIPTION:
The prevention of oral diseases is mainly targeted at the control of dental plaque. While tooth brushing is an effective method to remove plaque mechanically, it is not always sufficient and chemical antiplaque agents could be helpful. Some of them are used for their antibacterial action, the gold standard being chlorhexidine. Despite the great benefit of this bactericidal approach, the search continues for active ingredients that could prevent dental plaque formation without affecting the biological equilibrium within the oral cavity.

The aim of this study is to evaluate the efficiency of a mouthrinse, containing red grape seed extract and nicométhanol fluorhydrate, in the control of dental plaque deposit in a 4-days plaque regrowth model.

The study is a double blind randomized cross-over design, involving 50 healthy volunteers. During the treatment periods (4 days) no oral hygiene, measures excepting rinsing with the allocated product (active/non active) are permitted.

On day 1, the subjects receive professional prophylaxis. The mouthrinse is used pure, three times per day, after each meal. On day 5, subjects will be scored for disclosed plaque using the Quigley Hein index (modified by Turesky).

After a 2 weeks wash-out period, the subject receives the other product (active/non active) and uses it as in the first period.

On day 5, subjects will be scored again for disclosed plaque

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer
* without caries
* with at least 20 natural teeth excluding third molars
* Women using contraceptives for at least twelve weeks and while on study
* Protected by French social security system
* Written informed consent

Exclusion Criteria:

* Pregnancy or breast feeding
* Volunteers with partial denture or orthodontic appliance
* Person protected by the law who
* Person unable to give their consent to participate to the study.
* Under aged
* Current participation in another clinical trial
* Oral pathologies
* Systemic diseases
* Volunteers allergic to of the componentst of the tested products
* Volunteers with hyposalivation or xerostomia
* Treatment with antibiotics o intestinal antiseptics within 3 month before inclusion
* Treatment with oral antiseptics within 1 month before inclusion
* Alcoholic consumption more than 20 g/day (or 2 glasses)
* Heavy smokers
* Volunteers drinking a lot of tea or coffee

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-02; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Plaque index of Quickley-Hein modified by Tureski. Plaque deposits are scored on all natural teeth (except third molars) after staining. | Measures are done on days 5 of the two plaque growth periods

SECONDARY OUTCOMES:
Product tolerance | on days 5 of the two plaque growth periods
Product acceptability (oral sensation) | on days 5 of the two plaque growth periods

CONTACTS AND LOCATIONS:
Overall Officials: Cécile BADET, MD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux - Hôpital ST André - 1 rue Jean Burguet, Bordeaux, France

REFERENCES:
- [Background] Addy M. Evaluation of clinical trials of agents and procedures to prevent caries and periodontal disease: choosing products and recommending procedures. Int Dent J. 1995 Jun;45(3):185-96. PMID 7558357
- [Background] Guidelines for acceptance of chemotherapeutic products for the control of supragingival dental plaque and gingivitis. Council on Dental Therapeutics. J Am Dent Assoc. 1986 Apr;112(4):529-32. doi: 10.1016/s0002-8177(86)24021-0. No abstract available. PMID 3517110
- [Background] Yates RJ, Shearer BH, Morgan R, Addy M. A modification to the experimental gingivitis protocol to compare the antiplaque properties of two toothpastes. J Clin Periodontol. 2003 Feb;30(2):119-24. doi: 10.1034/j.1600-051x.2003.00205.x. PMID 12622853
- [Background] Furiga A, Lonvaud-Funel A, Dorignac G, Badet C. In vitro anti-bacterial and anti-adherence effects of natural polyphenolic compounds on oral bacteria. J Appl Microbiol. 2008 Nov;105(5):1470-6. doi: 10.1111/j.1365-2672.2008.03882.x. Epub 2008 Sep 13. PMID 18795979